CLINICAL TRIAL: NCT01051973
Title: Internet-delivered Cognitive Behavior Therapy Compared to Stress Management in the Treatment of Irritable Bowel Syndrome - A Randomized Controlled Study.
Brief Title: Cognitive Behavior Therapy (CBT) Compared to Stress Management for Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Brjann Ljotsson, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBS-X
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Cognitive behavior therapy; exposure; stress management
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavior therapy (Experimental)
  Interventions: Behavioral: Cognitive behavior therapy
- Stress management (Active Comparator)
  Interventions: Behavioral: Stress management

INTERVENTIONS:
Behavioral: Cognitive behavior therapy — A 10-week treatment based on exposure to symptoms and related feelings.
  Arms: Cognitive behavior therapy
Behavioral: Stress management — A 10-week stress management treatment including applied relaxation and dietary advice.
  Arms: Stress management

SUMMARY:
The study aims to compare two manualized treatments. They are based on cognitive behavior therapy or stress management. Both treatments are delivered via an internet application and the patients' work with the treatments is supported through online contact with a therapist. The treatments last for 10 weeks.

Approximately 200 patients will be included in the study and randomized to either condition.

The study hypothesis is that CBT will be superior to stress management on the main outcome measure, which is IBS symptom severity measured over 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBS given by physician
* At screening fulfilling Rome III-criteria for IBS

Exclusion Criteria:

* Severe depression
* Suicidal ideation
* Presence of unexplained IBS alarm symptoms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Level of IBS symptoms | During 4 consecutive weeks before randomization
  The Gastrointestinal symptom rating scale - IBS version. Mean of four weeks of assessment.
Level of IBS symptoms | During 4 consecutive weeks after treatment completion (10 weeks after randomization)
  The Gastrointestinal symptom rating scale - IBS version. Mean of four weeks of assessment.
Level of IBS symptoms | During 4 consecutive weeks 6 months after treatment completion
  The Gastrointestinal symptom rating scale - IBS version. Mean of four weeks of assessment.

SECONDARY OUTCOMES:
Quality of life | Before randomization, after treatment (10 weeks after randomization) and 6 months after treatment completion
  The Irritable Bowel Syndrome Quality of Life Instrument
Use of health care resources and societal production loss because of illness | Before randomization, after treatment (10 weeks after randomization) and 6 months after treatment completion
  Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry
Level of IBS-symptoms | Before randomization, after treatment (10 weeks after randomization) and 6 months after treatment completion
  IBS-Severity Scoring System
Anxiety related to gastrointestinal symptoms | Before randomization, after treatment (10 weeks after randomization) and 6 months after treatment completion
  Visceral Sensitivity Index
Level of daily stress | Before randomization, after treatment (10 weeks after randomization) and 6 months after treatment completion
  Perceived stress scale
Subjective relief of IBS-symptoms | Before randomization, after treatment (10 weeks after randomization) and 6 months after treatment completion
  One question: "In the past week, have you had adequate relief from IBS pain or discomfort?"

CONTACTS AND LOCATIONS:
Overall Officials: Nils Lindefors, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Internetpsykatrienheten, M57, Psykiatri sydväst, Stockholm, Sweden